CLINICAL TRIAL: NCT02977741
Title: Olanzapine for the Treatment of Refractory Chronic Nausea and Vomiting
Status: Withdrawn | Type: Observational
Why Stopped: Inability to recruit patients
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00037144
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Olanzapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Olanzapine

SUMMARY:
Prospective, observational study evaluating the effect of olanzapine for the treatment of refractory chronic nausea and vomiting.

DETAILED DESCRIPTION:
Patients will be identified who are seen in the Johns Hopkins Gastroenterology Clinic, suffer from chronic nausea and vomiting that is refractory to both prokinetic and antiemetic medications, and are being prescribed olanzapine for treatment of nausea and vomiting. Patients who meet criteria will be enrolled and their gastrointestinal symptoms, quality of life, and psychological symptoms will be assessed by various questionnaires and followed over the course of 3 months.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Able to communicate in English without aid of interpreter
* Have chronic refractory nausea, meeting each of the following criteria:

  1. Baseline nausea and vomiting score on VAS of 25mm or greater
  2. Duration symptoms of at least 6 months (does not have to be contiguous)
  3. Intolerance to or inadequate response to prior treatment with both 1) ondansetron or another serotonin (5HT3) antagonist and 2) metoclopramide or domperidone

Exclusion Criteria:

* History of chemotherapy within the last year
* Current diagnosis of cancer
* Pregnant or breastfeeding
* For females, active efforts to conceive/become pregnant during the time of the study
* Chronic opioid use (3 times a week or greater use)
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevation of greater than 2x upper limit of normal (within 3 months of enrollment)
* Cirrhosis
* Unable or unwilling to stop using metoclopramide while using olanzapine
* Concomitant use of other antipsychotics (e.g., haloperidol)
* Prolonged corrected QT interval (QTc) (>470ms for men and >480ms for women)
* History of life-threatening arrhythmia
* Hypokalemia (potassium <3.1) or hypomagnesemia (magnesium <1.2)
* Metabolic syndrome, defined as per Adult Treatment Panel III criteria
* Granulocytopenia (absolute neutrophil count <1500)
* History of tardive dyskinesia
* History of acute dystonic reaction to medications
* History of neuroleptic malignant syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who are seen in the Johns Hopkins Center for Neurogastroenterology, have been identified by the healthcare provider (physician, nurse practitioner, physician assistant) as having refractory chronic nausea and vomiting that has failed a trial of typical treatments (both anti-emetics and pro kinetics), and who will be prescribed olanzapine for the treatment of chronic nausea and vomiting
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Nausea and vomiting severity | 3 months
  Effect of olanzapine on refractory nausea and vomiting as per changes in patient scoring of the severity of nausea and vomiting on a daily visual analog scale (VAS). Scores range from 0-100, with higher scores indicating more severe symptoms.

SECONDARY OUTCOMES:
Severity of upper gastrointestinal symptoms | 3 months
  The effect of olanzapine on severity of upper gastrointestinal symptoms, assessed by the NIH Patient-Reported Outcomes Measurement Information System (PROMIS) Gastrointestinal Symptom Scales questionnaire. The questionnaire is 60-item GI symptom questionnaire covering 8 domains: Gastroesophageal reflux (13 items), disrupted swallowing (7 items), diarrhea (5 items), bowel incontinence/soilage (4 items), nausea and vomiting (4 items), constipation (9 items), belly pain (6 items), and gas/bloat/flatulence (12 items). Higher scores indicate more severe symptoms. A scoring service is used to convert the raw scores to a final T-score.
Quality of life and functional status | 3 months
  The effect of olanzapine on quality of life and functional status, assessed by the EuroQol 5 Dimension (EQ-5D) questionnaire. The EQ-5D descriptive system consists of five dimensions: Mobility, Self-care, Usual activities, Pain/discomfort, Anxiety/depression. Scores range from 5-25, with higher scores indicating more severe symptoms/decreased quality of life.
Symptom-specific anxiety | 3 months
  The effect of olanzapine on patient's overall gastrointestinal symptom-specific anxiety, assessed by the Visceral Sensitivity Index (VSI) questionnaire. The VSI is an instrument to assess gastrointestinal-specific anxiety, the cognitive, affective, and behavioral response to fear of gastrointestinal sensations, symptoms, and the context in which these visceral sensations and symptoms occur. The questionnaire consists of 15 questions, each scored 1-6. Total scores range from 15-90, with lower scores indicating more severe symptoms.
Presence of depression | 3 months
  Presence of depression in participants both before initiating olanzapine and after starting olanzapine, assessed by the Patient Health Questionnaire (PHQ-4) at baseline, 1 month, and 3 months. Total score is determined by adding together the scores for each of the 4 items. Scores range from 0-12 and are rated as normal (0-2), mild depression (3-5), moderate depression (6-8), and severe depression (9-12).

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States